CLINICAL TRIAL: NCT03184987
Title: A Phase III, 52-week, Open-label Study to Evaluate Long-term Safety of Fixed Dose Combination Therapy Fluticasone Furoate/Umeclidinium Bromide/Vilanterol Trifenatate in Japanese Patients With Asthma
Brief Title: A Long-term Safety Study of Fixed Dose Combination Therapy Fluticasone Furoate/Umeclidinium Bromide/Vilanterol Trifenatate in Japanese Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: York Bioanalytical Solution (Industry); BI Medical.Inc. (Industry); SRL Medisearch Inc. (Industry); Parexel (Industry); Q2 Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207236
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Results first posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: fluticasone furoate; fixed dose combination; Japanese subjects; vilanterol; asthma; umeclidinium bromide; closed triple therapy
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FF/UMEC/VI 100/62.5/25 mcg closed triple therapy (Experimental): Subjects will receive FF/UMEC/VI 100/62.5/25 mcg inhalation powder via ELLIPTA, once daily, 1 puff/time, in the morning. Subjects may receive salbutamol as a rescue medication when needed throughout the run-in and treatment period.
  Interventions: Drug: FF/UMEC/VI 100/62.5/25 mcg; Drug: Salbutamol; Other: ACQ-7
- FF/UMEC/VI 200/62.5/25 mcg closed triple therapy (Experimental): Subjects will receive FF/UMEC/VI 200/62.5/25 mcg inhalation powder via ELLIPTA, once daily, 1 puff/time, in the morning. Subjects may receive salbutamol as a rescue medication when needed throughout the run-in and treatment period.
  Interventions: Drug: FF/UMEC/VI 200/62.5/25 mcg; Drug: Salbutamol; Other: ACQ-7

INTERVENTIONS:
Drug: FF/UMEC/VI 100/62.5/25 mcg — Subjects will self-administer the study treatment via the ELLIPTA device. The ELLIPTA holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 100 mcg in each blister and the second strip contains UMEC 62.5 mcg and VI 25 mcg in each blister. ELLIPTA is a registered trademark of GSK groups of companies.
  Arms: FF/UMEC/VI 100/62.5/25 mcg closed triple therapy
Drug: FF/UMEC/VI 200/62.5/25 mcg — Subjects will self-administer the study treatment via the ELLIPTA device. The ELLIPTA holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 200 mcg in each blister and the second strip contains UMEC 62.5 mcg and VI 25 mcg in each blister. ELLIPTA is a registered trademark of GSK groups of companies.
  Arms: FF/UMEC/VI 200/62.5/25 mcg closed triple therapy
Drug: Salbutamol — Salbutamol is a rescue medication administered via metered-dose inhaler (MDI) which will be used when needed during the study.
Other: ACQ-7 — ACQ-7 will be used for the assessment of control status of asthma.

SUMMARY:
Despite availability of treatments and published guidelines, subjects may have asthma that is inadequately controlled. GlaxoSmithKline is currently developing a once-daily 'closed' triple therapy of an Inhaled Corticosteroids/Long-Acting Beta-2-Agonists/Long-Acting Muscarinic Antagonist (ICS/LAMA/LABA) combination (Fluticasone Furoate/Umeclidinium Bromide/Vilanterol Trifenatate [FF/UMEC/VI]) in a single device, with the aim of providing a new treatment option for the management of asthma by improving lung function, health-related quality of life (HRQoL) and symptom control over established combination therapies. This study has 3 study periods: Run-in, Treatment period and a Follow-up period. Eligible subjects who meet the pre-defined criteria at screening (Visit 1) will enter into a 2-week run-in period. Subjects will continue their pre-screening inhaled medications for asthma (ICS+LABA or ICS+LABA+LAMA) without any change in regimen/dosage until day before Visit 2. At Visit 2 subjects will be allocated to either FF/UMEC/VI 100/62.5/25 or FF/UMEC/VI 200/62.5/25 micrograms (mcg) treatment depending on the asthma control status for 52 weeks. Switching medication from FF/UMEC/VI 100/62.5/25 to FF/UMEC/VI 200/62.5/25 will be permitted in accordance with the control status of the subject assessed by Asthma Control Questionnaire (ACQ)-7 at Week 24 of the treatment period. A follow-up visit will be conducted for approximately 1 week. Subjects will be provided with salbutamol as a rescue medication throughout the study.

ELIGIBILITY:
Inclusion Criteria at the time of informed consent (Visit 0) and at screening (Visit 1).

* Age: Participant must be 18 years of age or older at the time of signing the informed consent.
* Ethnicity: Japanese
* Diagnosis: Subjects with a diagnosis of asthma as defined by the National Institutes of Health at least one year prior to providing informed consent.
* Current Asthma Maintenance Therapy: Outpatients are eligible if they have received ICS+LABA or ICS+LABA＋LAMA with asthma control status as Not well controlled with ICS (mid-dose) +LABA ; Not well controlled with ICS (high-dose) +LABA or Controlled with ICS (mid-dose) +LABA + LAMA; Not well controlled with ICS (mid-dose) +LABA + LAMA; Controlled with ICS (high-dose) +LABA + LAMA respectively in stable regimen and dosage for at least 4 weeks prior to screening visit (Visit 1) (with medium to high dose of ICS defined by the Japanese Guidelines [JGL]). Asthma Control Questionnaire (ACQ-6) will be used for the assessment of control status of asthma at Visit 1 (screening Visit) (i.e., less than or equal to 0.75 points shows controlled and > 0.75 shows not well controlled).
* Short-Acting Beta Agonists (SABAs): All subjects must be able to replace their current SABA inhaler with salbutamol aerosol inhaler at Visit 1 as needed for the duration of the study. Subjects should be able to withhold salbutamol for at least 6 hours prior to clinic visit.
* Sex: Male and/or female: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance from the screening visit until after the last dose of study medication and completion of the follow-up visit.
* Informed Consent: capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria at the time of informed consent (Visit 0) and at screening (Visit 1).

* Pneumonia: Chest X-ray documented pneumonia in the 6 weeks prior to Visit 1.
* Asthma Exacerbation: Any asthma exacerbation requiring a change in maintenance asthma therapy in the 6 weeks prior to Visit 1.
* COPD: Subjects with the diagnosis of chronic obstructive pulmonary disease, as per Global Initiative for Chronic Obstructive Lung Disease (GOLD 2016) guidelines, including history of exposure to risk factors (i.e., especially tobacco smoke, occupational dusts and chemicals, smoke from home cooking and heating fuels) (for tobacco smoke); post- salbutamol Forced Expiratory Volume in 1 second (FEV1)/forced vital capacity (FVC) ratio of <0.70 and a post- salbutamol FEV1 of less than or equal to 70% of predicted normal values (diagnosis prior to Visit 1 acceptable);Onset of disease greater than or equal to 40 years of age.
* Concurrent respiratory disorders: Subjects with current evidence of pneumonia, active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases or abnormalities other than asthma.
* Risk Factors for Pneumonia: Immune suppression (e.g., HIV, lupus) or other risk factors for pneumonia (e.g., neurological disorders affecting control of the upper airway, such as Parkinson's disease, myasthenia gravis). Patients at potentially high risk (e.g., very low body mass index (BMI), severely malnourished, or very low FEV1) will only be included at the discretion of the Investigator.
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).Note: Chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria.
* Clinically significant ECG abnormality: Evidence of a clinically significant abnormality in the 12-lead ECG performed during screening. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:

  * Atrial fibrillation (AF) with rapid ventricular rate >120 beats per minute (bpm)
  * Sustained or nonsustained ventricular tachycardia (VT)
  * Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted)
  * QT interval corrected for heart rate by Fridericia's formula (QTcF) greater than or equal to 500 milliseconds (msec) in patients with QRS <120 msec and QTcF greater than or equal to 530 msec in patients with QRS greater than or equal to 120 msec.
* Unstable or life threatening cardiac disease: subjects with any of the following at screening (Visit 1) would be excluded:

  * Myocardial infarction or unstable angina in the last 6 months
  * Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months
  * New York Heart Association (NYHA) Class IV heart failure
* Antimuscarinic effects: Subjects with a medical condition such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction should only be included if in the opinion of the Investigator the benefit outweighs the risk and that the condition would not contraindicate study participation.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the subject has been considered cured by treatment.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Medication prior to spirometry: Subjects who are medically unable to withhold their salbutamol for the 6-hour period required prior to spirometry testing at each study visit.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Allergy or hypersensitivity: A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta-agonist, lactose/severe milk protein or magnesium stearate.
* Tobacco use: Subjects who are: Current smokers (defined as subjects who have used inhaled tobacco products within the 12 months prior to Visit 1 [i.e., cigarettes, e-cigarettes/vaping, cigars or pipe tobacco]); Former smokers with a smoking history of greater than equal to 10 pack years (e.g., greater than equal to 20 cigarettes/day for 10 years).
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Affiliation with Investigator site: Study Investigators, sub-Investigators, study coordinators, employees of a participating Investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* Inability to read: In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials.

Inclusion Criteria end of the run-in period (Visit 2)

* Asthma maintenance therapy: No changes in asthma maintenance therapy (excluding salbutamol inhalation aerosol provided at Visit 1) and control status during the run-in period. Asthma Control Questionnaire (ACQ-6 at screening and ACQ-7 at the end of the run-in period) will be used for the assessment of control status of asthma, i.e., 0.75 points shows controlled and >0.75 shows not well controlled.
* Concurrent conditions/medical history: Liver function test at Visit1

  * ALT <2 x upper limit of normal (ULN)
  * ALP less than or equal to 1.5 x ULN
  * Bilirubin less than or equal to 1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)

Exclusion Criteria end of the run-in period (Visit 2)

* Respiratory Infection: Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Severe asthma exacerbation: Evidence of a severe exacerbation during screening or the run-in period, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
* Laboratory test abnormalities: Evidence of clinically significant abnormal laboratory tests during screening or the run-in period which are still abnormal upon repeat analysis and are not believed to be due to disease(s) present. Each Investigator will use his/her own discretion in determining the clinical significance of the abnormality.
* There is no restriction on diet in this study.
* Use of tobacco products will not be allowed from screening until after the final follow-up visit. Caffeine and alcohol is allowed ad libitum.
* There is no restriction on activity in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated long-term safety of fixed dose combination therapy Fluticasone Furoate/Umeclidinium Bromide/Vilanterol Trifenatate (FF/UMEC/VI) in Japanese participants with asthma. The study was conducted across multiple centers in Japan.
Pre-assignment Details: A total of 114 participants were screened, of which 1 failed screening and 2 participants were run-in failures and 111 participants received study treatment.
Groups:
- FF/UMEC/VI 100/62.5/25 mcg: Participants received FF/UMEC/VI 100/62.5/25 microgram (mcg) inhalation powder via ELLIPTA, once daily in the morning for 52 weeks. Participants received salbutamol via metered-dose inhaler as a rescue medication during the study.
- FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg: Participants were administered FF/UMEC/VI 100/62.5/25 mcg via ELLIPTA once daily in the morning for 24 weeks. Participants with inadequate asthma control as assessed by Asthma Control Questionnaire-7 (ACQ-7) (i.e. ACQ score >0.75) could be switched treatment from FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg at Week 24 of the treatment period based on the ACQ-7. Participants were administered salbutamol via metered-dose inhaler as a rescue medication.
- FF/UMEC/VI 200/62.5/25 mcg: Participants received FF/UMEC/VI 200/62.5/25 mcg inhalation powder via ELLIPTA once daily in the morning for 52 weeks. Participants were administered salbutamol via metered-dose inhaler as a rescue medication.
Period: Overall Study
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Started | 47 | 9 | 55
Completed | 46 | 8 | 51
Not Completed | 1 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FF/UMEC/VI 100/62.5/25 mcg: Participants received FF/UMEC/VI 100/62.5/25 mcg inhalation powder via ELLIPTA once daily in the morning for 52 weeks. Participants received salbutamol via metered-dose inhaler as a rescue medication during the study.
- Total: Total of all reporting groups
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg | Total
Number analyzed (Participants) | 47 | 9 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (14.28) | 48.4 (7.76) | 53.8 (12.91) | 50.9 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 5 | 36 | 64
  Male | 24 | 4 | 19 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Japanese/East Asian Heritage (EAH)/South EAH | 47 | 9 | 55 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose: result in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect, other important medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the outcome mentioned before. Intent-To-Treat (ITT) Population comprised of all participants who received at least one dose of study treatment in the treatment period.
Time Frame: Up to Week 52
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Participants
  Non-SAEs | 23 | 7 | 32
  SAEs | 1 | 0 | 2

2. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in seated position after 5 minutes rest for participants at indicated time points. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 4, 12, 24, 36 and 52
Population: ITT Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Millimeters of mercury
  SBP: Week 4, n=47,9,55 | -1.9 (11.27) | 7.4 (9.91) | 2.7 (12.66)
  SBP: Week 12, n=47,9,55 | -1.7 (10.35) | 1.2 (12.25) | 4.6 (12.10)
  SBP: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  SBP: Week 24, n=46,9,52 | -0.9 (11.68) | -1.0 (13.87) | 3.3 (12.85)
  SBP: Week 36, n=46,8,52: number analyzed (Participants) | 46 | 8 | 52
  SBP: Week 36, n=46,8,52 | 2.0 (12.60) | 5.0 (15.92) | 4.6 (12.62)
  SBP: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  SBP: Week 52, n=46,8,51 | 0.1 (9.21) | 3.6 (9.07) | 3.4 (13.09)
  DBP: Week 4, n=47,9,55 | 1.6 (6.04) | 3.3 (4.64) | -0.2 (7.63)
  DBP: Week 12, n=47,9,55 | -0.1 (9.07) | -0.2 (7.76) | 1.7 (8.66)
  DBP: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  DBP: Week 24, n=46,9,52 | 0.4 (8.32) | 1.6 (5.75) | 2.1 (8.22)
  DBP: Week 36, n=46,8,52: number analyzed (Participants) | 46 | 8 | 52
  DBP: Week 36, n=46,8,52 | 4.2 (7.18) | 4.8 (7.40) | 3.1 (9.93)
  DBP: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  DBP: Week 52, n=46,8,51 | 2.1 (6.98) | 2.4 (3.70) | 2.5 (9.60)

3. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in seated position after 5 minutes rest for participants at indicated time points. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 4, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Beats per minute
  Week 4, n=47,9,55 | 0.3 (9.28) | 5.9 (7.04) | 1.6 (7.85)
  Week 12, n=47,9,55 | -0.1 (9.58) | 4.4 (7.14) | 2.3 (7.55)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -2.6 (8.63) | 4.6 (7.73) | -1.8 (6.35)
  Week 36, n=46,8,52: number analyzed (Participants) | 46 | 8 | 52
  Week 36, n=46,8,52 | 2.4 (11.65) | 7.0 (9.27) | 4.2 (8.41)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -0.3 (8.94) | -1.4 (2.45) | 1.7 (9.22)

4. Secondary Outcome: Change From Baseline in PR Interval and QT Interval Corrected for Heart Rate According to Fridericia's Formula (QTcF)
Description: Single 12-lead electrocardiograms (ECG) were obtained using an automated ECG machine that measured PR Interval and QTcF Interval. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 4, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Milliseconds
  PR Interval: Week 4, n=47,9,55 | -2.3 (10.12) | 5.1 (10.62) | -0.3 (9.40)
  PR Interval: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  PR Interval: Week 24, n=46,9,52 | 1.5 (9.43) | -0.4 (12.12) | 2.5 (10.29)
  PR Interval: Week 52, n=46,8,50: number analyzed (Participants) | 46 | 8 | 50
  PR Interval: Week 52, n=46,8,50 | -1.3 (10.11) | 1.3 (9.57) | 1.7 (8.97)
  QTcF Interval: Week 4, n=47,9,55 | -1.890 (11.3898) | 1.757 (13.8084) | 3.914 (27.5206)
  QTcF Interval: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  QTcF Interval: Week 24, n=46,9,52 | -1.577 (10.4434) | 7.578 (8.0630) | -3.265 (14.3663)
  QTcF Interval: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  QTcF Interval: Week 52, n=46,8,51 | 1.745 (13.3558) | 3.243 (17.5127) | 0.969 (15.3699)

5. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Picograms
  Week 12, n=47,9,55 | -0.04 (0.591) | 0.49 (1.190) | 0.09 (0.803)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | 0.41 (0.674) | 0.76 (1.254) | 0.35 (0.764)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | 0.07 (0.915) | 0.66 (1.571) | 0.22 (0.833)

6. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Femtoliters
  Week 12, n=47,9,55 | -0.55 (1.525) | 0.90 (3.240) | -0.20 (2.112)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | 0.35 (1.499) | 1.49 (2.336) | 0.69 (2.208)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | 0.21 (1.978) | 1.76 (2.753) | 0.55 (2.707)

7. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
10^12 cells per liter
  Week 12, n=47,9,55 | -0.084 (0.2046) | -0.161 (0.2421) | -0.056 (0.1868)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -0.123 (0.1908) | -0.109 (0.2158) | -0.101 (0.2114)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -0.024 (0.1905) | -0.055 (0.2321) | -0.032 (0.2026)

8. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Percentage of red blood cells in blood
  Week 12, n=47,9,55 | -0.0102 (0.01714) | -0.0103 (0.02148) | -0.0061 (0.01616)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -0.0100 (0.01627) | -0.0029 (0.01527) | -0.0063 (0.01878)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -0.0011 (0.01602) | 0.0034 (0.02251) | 0.0001 (0.01749)

9. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Grams per liter
  Week 12, n=47,9,55 | -2.6 (6.19) | -2.4 (7.92) | -1.3 (5.66)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -2.0 (6.33) | 0.2 (6.20) | -1.5 (5.77)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -0.4 (6.47) | 1.4 (9.32) | 0.3 (6.01)

10. Secondary Outcome: Change From Baseline in Hematology Parameter: Platelet Count
Description: Blood samples were collected to analyze the hematology parameter: platelet count. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
10^9 cells per liter
  Week 12, n=47,9,55 | 3.8 (27.46) | -17.7 (37.26) | 4.8 (33.99)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | 3.1 (28.67) | -20.6 (54.69) | 4.6 (39.72)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -2.8 (27.48) | -18.4 (51.83) | 3.3 (25.73)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Basophils/Leukocytes
Description: Blood samples were collected to analyze the hematology parameter: Basophils/Leukocytes. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of basophil in leukocytes
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Percentage of basophil in leukocytes
  Week 12, n=47,9,55 | 0.01 (0.352) | -0.03 (0.600) | -0.10 (0.440)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | 0.02 (0.334) | -0.03 (0.487) | -0.05 (0.365)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | 0.10 (0.373) | 0.01 (0.295) | 0.05 (0.363)

12. Secondary Outcome: Change From Baseline in Hematology Parameter: Eosinophils/Leukocytes
Description: Blood samples were collected to analyze the hematology parameter: Eosinophils/Leukocytes. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils in leukocytes
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Percentage of eosinophils in leukocytes
  Week 12, n=47,9,55 | -0.35 (2.140) | -0.18 (3.500) | -0.87 (3.553)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -0.13 (2.694) | 1.68 (2.859) | 0.19 (3.015)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | 0.58 (2.924) | 0.01 (5.046) | 0.13 (4.371)

13. Secondary Outcome: Change From Baseline in Hematology Parameter: Lymphocytes/Leukocytes
Description: Blood samples were collected to analyze the hematology parameter: Lymphocytes/Leukocytes. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes in leukocytes
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Percentage of lymphocytes in leukocytes
  Week 12, n=47,9,55 | -1.77 (7.644) | -0.12 (6.009) | -0.95 (6.324)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -0.75 (5.431) | -3.20 (6.279) | -2.06 (5.282)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -0.26 (5.198) | -0.07 (7.054) | -1.54 (5.672)

14. Secondary Outcome: Change From Baseline in Hematology Parameter: Monocytes/Leukocytes
Description: Blood samples were collected to analyze the hematology parameter: Monocytes/Leukocytes. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of monocytes in leukocytes
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Percentage of monocytes in leukocytes
  Week 12, n=47,9,55 | -0.48 (1.717) | 0.03 (1.141) | -0.34 (1.229)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | -0.49 (1.518) | 0.20 (1.683) | 0.17 (1.468)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | 0.14 (1.400) | -0.19 (1.174) | -0.04 (1.009)

15. Secondary Outcome: Change From Baseline in Hematology Parameter: Neutrophils/Leukocytes
Description: Blood samples were collected to analyze the hematology parameter: Neutrophils/Leukocytes. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils in leukocytes
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Percentage of neutrophils in leukocytes
  Week 12, n=47,9,55 | 2.59 (8.777) | 0.30 (7.925) | 2.26 (8.081)
  Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Week 24, n=46,9,52 | 1.36 (6.599) | 1.36 (9.352) | 1.76 (7.257)
  Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Week 52, n=46,8,51 | -0.56 (6.487) | 0.24 (8.451) | 1.40 (7.512)

16. Secondary Outcome: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase
Description: Blood samples were collected to analyze the chemistry parameters: alanine aminotransferase, alkaline phosphatase and aspartate aminotransferase. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
International units per liter
  Alanine aminotransferase: Week 12, n=47,9,55 | -0.0 (8.56) | -2.1 (6.51) | -1.5 (10.23)
  Alanine aminotransferase: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Alanine aminotransferase: Week 24, n=46,9,52 | -1.5 (8.62) | -0.4 (4.50) | 0.3 (13.91)
  Alanine aminotransferase: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Alanine aminotransferase: Week 52, n=46,8,51 | -2.3 (10.07) | -1.1 (4.49) | 1.4 (22.10)
  Alkaline phosphatase: Week 12, n=47,9,55 | 1.0 (22.83) | 2.0 (14.56) | -13.2 (36.95)
  Alkaline phosphatase: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Alkaline phosphatase: Week 24, n=46,9,52 | -4.3 (20.89) | 2.6 (30.69) | -8.1 (41.91)
  Alkaline phosphatase: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Alkaline phosphatase: Week 52, n=46,8,51 | 2.3 (26.70) | -7.9 (31.86) | -7.2 (38.89)
  Aspartate aminotransferase: Week 12, n=47,9,55 | -0.4 (8.05) | -0.6 (2.70) | -1.3 (6.44)
  Aspartate aminotransferase: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Aspartate aminotransferase: Week 24, n=46,9,52 | -2.0 (8.10) | 0.6 (2.46) | -0.0 (9.37)
  Aspartate aminotransferase: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Aspartate aminotransferase: Week 52, n=46,8,51 | -2.1 (9.80) | 0.3 (3.15) | 0.6 (11.36)

17. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin and protein. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Grams per liter
  Albumin: Week 12, n=47,9,55 | 0.2 (2.60) | 0.4 (4.10) | 0.1 (2.27)
  Albumin: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Albumin: Week 24, n=46,9,52 | -0.3 (2.02) | -0.1 (5.53) | -0.3 (2.24)
  Albumin: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Albumin: Week 52, n=46,8,51 | -0.2 (2.27) | -0.9 (3.80) | -0.6 (1.93)
  Protein: Week 12, n=47,9,55 | -0.2 (3.06) | -0.1 (3.79) | -0.1 (3.43)
  Protein: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Protein: Week 24, n=46,9,52 | -1.4 (2.59) | -0.7 (3.71) | -0.8 (3.10)
  Protein: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Protein: Week 52, n=46,8,51 | -0.6 (3.12) | -1.4 (4.07) | -0.7 (3.17)

18. Secondary Outcome: Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: bilirubin, creatinine and direct bilirubin. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Micromoles per liter
  Bilirubin: Week 12, n=47,9,55 | 0.764 (3.5263) | 2.850 (2.7037) | 1.213 (3.0103)
  Bilirubin: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Bilirubin: Week 24, n=46,9,52 | 0.967 (2.8535) | 3.040 (3.8024) | -0.230 (4.0214)
  Bilirubin: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Bilirubin: Week 52, n=46,8,51 | 0.223 (3.0718) | 2.779 (1.8137) | 0.000 (3.2445)
  Creatinine: Week 12, n=47,9,55 | 0.3762 (5.16031) | 0.3929 (7.64431) | 1.2697 (6.83001)
  Creatinine: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Creatinine: Week 24, n=46,9,52 | 2.1139 (4.90769) | -0.4911 (5.04173) | 0.9860 (5.01490)
  Creatinine: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Creatinine: Week 52, n=46,8,51 | 0.6918 (4.88441) | -0.7735 (4.85194) | 0.9533 (5.52579)
  Direct bilirubin: Week 12, n=47,9,55 | 0.182 (1.4366) | 0.950 (0.9012) | 0.155 (1.2433)
  Direct bilirubin: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Direct bilirubin: Week 24, n=46,9,52 | 0.149 (0.8701) | 1.140 (1.2092) | -0.329 (1.3561)
  Direct bilirubin: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Direct bilirubin: Week 52, n=46,8,51 | -0.223 (1.3299) | 0.641 (0.8850) | -0.101 (1.1035)

19. Secondary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: calcium, glucose, potassium, sodium and urea. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as relevant visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Millimoles per liter
  Calcium: Week 12, n=47,9,55 | 0.0021 (0.07464) | -0.0083 (0.08461) | -0.0245 (0.23525)
  Calcium: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Calcium: Week 24, n=46,9,52 | -0.0016 (0.06805) | -0.0055 (0.12399) | 0.0043 (0.07586)
  Calcium: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Calcium: Week 52, n=46,8,51 | 0.0125 (0.07815) | 0.0000 (0.09335) | 0.0313 (0.06560)
  Glucose: Week 12, n=47,9,55 | 0.0343 (0.90775) | -0.0370 (0.58286) | 0.1605 (0.82194)
  Glucose: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Glucose: Week 24, n=46,9,52 | 0.1255 (0.68761) | 0.0247 (0.40136) | 0.2701 (0.79361)
  Glucose: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Glucose: Week 52, n=46,8,51 | 0.0567 (0.78708) | 0.1804 (0.46514) | 0.1099 (0.66570)
  Potassium: Week 12, n=47,9,55 | -0.01 (0.326) | -0.07 (0.206) | -0.04 (0.301)
  Potassium: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Potassium: Week 24, n=46,9,52 | -0.01 (0.308) | 0.07 (0.357) | -0.06 (0.306)
  Potassium: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Potassium: Week 52, n=46,8,51 | 0.03 (0.293) | 0.04 (0.346) | 0.03 (0.300)
  Sodium: Week 12, n=47,9,55 | -0.2 (1.77) | -0.3 (2.00) | -0.1 (2.13)
  Sodium: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Sodium: Week 24, n=46,9,52 | -0.5 (1.81) | -1.0 (1.80) | -0.3 (1.89)
  Sodium: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Sodium: Week 52, n=46,8,51 | -0.4 (2.13) | -0.8 (1.83) | -0.2 (2.28)
  Urea: Week 12, n=47,9,55 | -0.1162 (1.16663) | -0.9282 (1.68737) | 0.1889 (1.26748)
  Urea: Week 24, n=46,9,52: number analyzed (Participants) | 46 | 9 | 52
  Urea: Week 24, n=46,9,52 | -0.5301 (1.16959) | -1.3328 (1.64540) | -0.2018 (1.01357)
  Urea: Week 52, n=46,8,51: number analyzed (Participants) | 46 | 8 | 51
  Urea: Week 52, n=46,8,51 | -0.2398 (1.50149) | -0.4641 (1.28392) | -0.0224 (1.17972)

20. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Urinalysis Results Relative to Baseline
Description: Urine samples were collected for analysis of presence of occult blood and protein in urine using dipstick method. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of occult blood and protein can be read as Trace, 1+, 2+ and 3+ indicating proportional concentrations in the urine sample. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to Week 52
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 47 | 9 | 55
Participants
  Occult Blood; No Change/Decreased | 39 | 7 | 44
  Occult Blood; Increase to Trace | 1 | 0 | 0
  Occult Blood; Increase to 1+ | 2 | 0 | 4
  Occult Blood; Increase to 2+ | 2 | 1 | 3
  Occult Blood; Increase to 3+ | 3 | 1 | 4
  Protein; No Change/Decreased | 32 | 7 | 34
  Protein; Increase to Trace | 10 | 1 | 14
  Protein; Increase to 1+ | 5 | 0 | 5
  Protein; Increase to 2+ | 0 | 1 | 2
  Protein; Increase to 3+ | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from Day 1 up to Week 52
Description: ITT Population comprised of all participants who received at least one dose of study treatment in the treatment period.
Arm/Group | FF/UMEC/VI 100/62.5/25 mcg | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/9 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/9 | 2/55
Other Adverse Events (participants affected / at risk) | 23/47 | 7/9 | 32/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/UMEC/VI 100/62.5/25 mcg (N=47) | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg (N=9) | FF/UMEC/VI 200/62.5/25 mcg (N=55)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/UMEC/VI 100/62.5/25 mcg (N=47) | FF/UMEC/VI 100/62.5/25 mcg to FF/UMEC/VI 200/62.5/25 mcg (N=9) | FF/UMEC/VI 200/62.5/25 mcg (N=55)
Nasopharyngitis (Infections and infestations) | 13 | 2 | 18
Pharyngitis (Infections and infestations) | 5 | 2 | 4
Bronchitis (Infections and infestations) | 4 | 2 | 4
Influenza (Infections and infestations) | 3 | 1 | 5
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Rhinitis (Infections and infestations) | 2 | 0 | 3
Acute sinusitis (Infections and infestations) | 1 | 1 | 2
Chronic sinusitis (Infections and infestations) | 1 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Eustachian tube stenosis (Ear and labyrinth disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03184987/SAP_000.pdf
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03184987/Prot_001.pdf